CLINICAL TRIAL: NCT01298063
Title: Pharmacokinetics, Safety and Tolerability of Different Oral Doses of Afatinib, in Subjects With Mild to Moderate Hepatic Impairment Compared to Healthy Subjects - a Phase I, Single-dose, Open-label, Dose-escalation Study in a Matched Group Design
Brief Title: Influence of Mild and Moderate Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of Various Doses of Afatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.86; 2010-021140-18 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-08

CONDITIONS: Liver Diseases; Healthy
MeSH Terms: conditions — Liver Diseases | interventions — Afatinib

ARMS (3):
- Afatinib Group A, B (2), D (Experimental): healthy subjects, mild and moderate liver impaired subjects to receive one single dose treatment containing the highest dose afatinib
  Interventions: Drug: Afatinib
- Afatinib Group B (3), D (Experimental): healthy subjects, moderate liver impaired subjects to receive one single dose treatment containing the medium dose of afatinib
  Interventions: Drug: Afatinib
- Afatinib Group B (1), D (Experimental): healthy subjects, moderate liver impaired subjects to receive one single dose treatment containing the low dose of afatinib
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — 1 tablet, once qd in the morning
  Arms: Afatinib Group A, B (2), D
Drug: Afatinib — 1 tablet, once qd in the morning
  Arms: Afatinib Group B (3), D
Drug: Afatinib — 1 tablet, once qd in the morning
  Arms: Afatinib Group B (1), D

SUMMARY:
Up to 38 subjects entered with the aim of entering 8 subjects with mild liver impairment (at highest dose of afatinib), 8 subjects with moderate liver impairment (at either highest dose or two lower doses) and 8 healthy matched controls to each of this two groups.

ELIGIBILITY:
Inclusion criteria:

Healthy subjects:

1. Healthy males and females according to a complete medical history, including a physical examination, vital signs (Blood Pressure, Pulse Rate), 12-lead Electrocardiogram, and clinical laboratory tests. The healthy subjects must meet the matching criteria based on the matching approach (cf. Section 3.3).
2. Age =18 and =75 years
3. Body Mass Index =18.5 and =34 kg/m2
4. Creatinine clearance >70 mL/min according to Cockroft & Gault (for healthy volunteers, cf. Section 10.2)
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation. Hepatically impaired subjects as determined by a hepatologist/ gastroenterologist:
6. Male and female liver impaired subjects determined by results of screening classified as Child-Pugh A; Child-Pugh score of 5-6 points or as Child-Pugh B; Child-Pugh score of 7-9 points, cf. Section 10.2. Child-Pugh criteria must be stable for at least 3 months prior to screening and during the trial.
7. Age =18 and =75 years
8. Body Mass Index =18.5 and =34 kg/m2
9. Creatinine clearance >40 mL/min according to Cockroft & Gault (for liver impaired subjects, cf. Section 10.2)
10. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation.

    For all females:
11. Postmenopausal female subjects (postmenopausal defined as at least 1 year of spontaneous amenorrhea [in questionable cases or spontaneous amenorrhea below 1 year a blood sample with simultaneous follicle stimulating hormone (FSH) above 40 IU/l and estradiol below 30 ng/l is confirmatory]) or adequate contraception* for female subjects of childbearing potential during the study and until 2 months after study completion, e.g. any of the following: implants, injectables, combined oral contraceptives, IUD (intrauterine device), sexual abstinence for at least 1 month prior to first study drug administration, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who do not have a vasectomised partner, are not sexually abstinent or surgically sterile have to use an additional barrier method (e.g. condom).

Exclusion criteria:

Any relevant deviation from healthy conditions (excluded conditions caused by liver impairment)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1200.86.1 Boehringer Ingelheim Investigational Site, Kiel, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 mg Afatinib Group A: Group A: Mild hepatic impaired subjects with Child Pugh A were treated with 50 milligram (mg) Afatinib (One tablet qd in the morning).
- 30 mg Afatinib Group B1: Group B1: Moderate hepatic impaired subjects with Child Pugh B were treated with 30 mg Afatinib (One tablet qd in the morning).
- 50 mg Afatinib Group B2: Group B2: Moderate hepatic impaired subjects with Child Pugh B were treated with 50 mg Afatinib (One tablet qd in the morning).
- 50 mg Afatinib Group C: Group C: Subjects with normal hepatic function matching to subjects in group A were treated with 50 mg Afatinib (One tablet qd in the morning).
- 50 mg Afatinib Group D: Group D: Subjects with normal hepatic function matching to subjects in group B2 were treated with 50 mg Afatinib (One tablet qd in the morning).
Period: Overall Study
Arm/Group | 50 mg Afatinib Group A | 30 mg Afatinib Group B1 | 50 mg Afatinib Group B2 | 50 mg Afatinib Group C | 50 mg Afatinib Group D
Started | 8 | 3 | 8 | 8 | 8
Completed | 8 | 3 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 50 mg Afatinib Group A: Group A: Mild hepatic impaired subjects with Child Pugh A were treated with 50 mg Afatinib (One tablet qd in the morning).
- Total: Total of all reporting groups
Arm/Group | 50 mg Afatinib Group A | 30 mg Afatinib Group B1 | 50 mg Afatinib Group B2 | 50 mg Afatinib Group C | 50 mg Afatinib Group D | Total
Number analyzed (Participants) | 8 | 3 | 8 | 8 | 8 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (9.0) | 64.3 (6.1) | 54.8 (9.0) | 55.9 (12.6) | 53.1 (7.9) | 55.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 2 | 3 | 10
  Male | 6 | 3 | 5 | 6 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve From 0 to Infinity (AUC0-infinity)
Description: AUC0-infinity represents the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity
Time Frame: 30 minutes (min) prior to first dosing and 30 min, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 9 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 h, 240 h after first dosing
Population: Pharmacokinetic (PK) analysis set includes all evaluable matched subjects in the treated set providing at least 1 observation for at least 1 PK endpoint without important protocol violations. Group B1 was not included in the primary analysis set for comparison.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 50 mg Afatinib Group A | 30 mg Afatinib Group B1 | 50 mg Afatinib Group B2 | 50 mg Afatinib Group C | 50 mg Afatinib Group D
Number analyzed (Participants) | 8 | 3 | 8 | 8 | 8
ng*h/mL | 886 (53.7) | 552 (42.1) | 934 (31.0) | 956 (22.7) | 985 (32.3)
Statistical Analysis 1: Comparison: 50 mg Afatinib Group A vs 50 mg Afatinib Group C; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.1998, ANOVA — P-value for ratio outside interval 80 - 125 percent; Adjusted (by treatment) geometric mean ratio; Geometric mean ratio = 92.64, 90% CI 2-sided [67.960 to 126.270], Standard Deviation 33.6 — The standard deviation is actually the intra individual geometric coefficient of variation
Statistical Analysis 2: Comparison: 50 mg Afatinib Group B2 vs 50 mg Afatinib Group D; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.1440, ANOVA — P-value for ratio outside interval 80 - 125 percent; Adjusted (by treatment) geometric mean ratio; Geometric mean ratio = 94.88, 90% CI 2-sided [72.278 to 124.549], Standard Deviation 31.6 — The standard deviation is actually the intra individual geometric coefficient of variation

2. Primary Outcome: Maximum Concentration (Cmax)
Description: Cmax represents the maximum measured concentration of the analyte in plasma
Time Frame: as for outcome 1
Population: PK analysis set. Group B1 was not included in the primary analysis set for comparison.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 50 mg Afatinib Group A | 30 mg Afatinib Group B1 | 50 mg Afatinib Group B2 | 50 mg Afatinib Group C | 50 mg Afatinib Group D
Number analyzed (Participants) | 8 | 3 | 8 | 8 | 8
ng/mL | 33.7 (51.7) | 17.5 (44.1) | 39.5 (40.1) | 30.7 (33.7) | 31.1 (46.0)
Statistical Analysis 1: Comparison: 50 mg Afatinib Group A vs 50 mg Afatinib Group C; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.2002, ANOVA — P-value for ratio outside interval 80 - 125 percent; Adjusted (by treatment) geometric mean ratio; Geometric mean ratio = 109.47, 90% CI 2-sided [82.683 to 144.947], Standard Deviation 30.3 — The standard deviation is actually the intra individual geometric coefficient of variation
Statistical Analysis 2: Comparison: 50 mg Afatinib Group B2 vs 50 mg Afatinib Group D; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.5281, ANOVA — P-value for ratio outside interval 80 - 125 percent; Adjusted (by treatment) geometric mean ratio; Geometric mean ratio = 126.89, 90% CI 2-sided [86.028 to 187.159], Standard Deviation 42.8 — The standard deviation is actually the intra individual geometric coefficient of variation

3. Secondary Outcome: Area Under Curve From 0 to tz (AUC0-tz)
Description: AUC0-tz represents the area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point
Time Frame: as for outcome 1
Population: PK analysis set. Group B1 was not included in the primary analysis set for comparison.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 50 mg Afatinib Group A | 30 mg Afatinib Group B1 | 50 mg Afatinib Group B2 | 50 mg Afatinib Group C | 50 mg Afatinib Group D
Number analyzed (Participants) | 8 | 3 | 8 | 8 | 8
ng*h/mL | 842 (50.8) | 519 (39.1) | 904 (31.4) | 930 (22.5) | 956 (33.3)
Statistical Analysis 1: Comparison: 50 mg Afatinib Group A vs 50 mg Afatinib Group C; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.2309, ANOVA — P-value for ratio outside interval 80 - 125 percent; Adjusted (by treatment) geometric mean ratio; Geometric mean ratio = 90.61, 90% CI 2-sided [66.915 to 122.705], Standard Deviation 32.8 — The standard deviation is actually the intra individual geometric coefficient of variation
Statistical Analysis 2: Comparison: 50 mg Afatinib Group B2 vs 50 mg Afatinib Group D; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.1546, ANOVA — P-value for ratio outside interval 80 - 125 percent; Adjusted (by treatment) geometric mean ratio; Geometric mean ratio = 94.49, 90% CI 2-sided [71.563 to 124.764], Standard Deviation 32.4 — The standard deviation is actually the intra individual geometric coefficient of variation

4. Secondary Outcome: Clinical Relevant Abnormalitites for Physical Examination, Vital Signs, 12-lead ECG, Clinical Laboratory Tests, Adverse Event, Investigator's Global Tolerability
Description: Clinical relevant abnormalitites for physical examination, vital signs, 12-lead electrocardiogramm (ECG), clinical laboratory test (including hematology, clinical chemistry, coagulation, urinalysis), adverse event, investigator's global tolerability. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Population: Treated set
Measure: Number; unit: participants
Arm/Group | 50 mg Afatinib Group A | 30 mg Afatinib Group B1 | 50 mg Afatinib Group B2 | 50 mg Afatinib Group C | 50 mg Afatinib Group D
Number analyzed (Participants) | 8 | 3 | 8 | 8 | 8
participants
  Lipase increased | 1 | 0 | 0 | 0 | 0
  Hyperlipasaemia | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | 50 mg Afatinib Group A | 30 mg Afatinib Group B1 | 50 mg Afatinib Group B2 | 50 mg Afatinib Group C | 50 mg Afatinib Group D
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 1/3 | 1/8 | 1/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Afatinib Group A (N=8) | 30 mg Afatinib Group B1 (N=3) | 50 mg Afatinib Group B2 (N=8) | 50 mg Afatinib Group C (N=8) | 50 mg Afatinib Group D (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.